CLINICAL TRIAL: NCT07354568
Title: Prognosis of Patients With Mixed Cardiogenic-Vasoplegic Shock: a French Multicenter Cohort
Brief Title: Prognosis of Patients With Mixed Cardiogenic-Vasoplegic Shock
Acronym: PROMIX
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, Beyls, Doctor, Principal Investigator, Centre Hospitalier Universitaire, Amiens
Other Study IDs: PI2025_843_0187; N° HDH : 27130053 (Other: Health Data Hub)
Record Dates: First submitted 2025-12-15; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiogenic Shock Acute; Bypass, Cardiopulmonary; Septic Shock; Mechanical Circulatory Support; Myocardial Infarction (MI); Cardiogenic Shock Post Myocardial Infarction
Keywords: VA-ECMO; Cardiogenic Shock; Mechanical Circulatory Support; Vasopressor; Mixed Cardiogenic Shock; post cardiotomy shock
MeSH Terms: conditions — Shock, Septic; Myocardial Infarction; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Mixed Cardiogenic-Vasoplegia Shock: Patients hospitalized in an intensive care unit (ICU) or cardiac ICU for cardiogenic shock, at least stage C according to the SCAI classification.
  Vasoplegia was defined by the requirement of norepinephrine > 0.20 µg/kg/min (γ/kg/min) to maintain a mean arterial pressure ≥ 65 mmHg.
- Patients with Cardiogenick Shock Without Vasoplegia: Patients hospitalized in an intensive care unit (ICU) or cardiac ICU for cardiogenic shock, at least stage C according to the SCAI classification.

SUMMARY:
Mixed cardiogenic-vasoplegic shock (M-CS) represents a distinct and severe phenotype of cardiogenic shock characterized by concomitant myocardial dysfunction and inappropriate systemic vasodilation. Despite its clinical relevance, the epidemiology, management, and outcomes of M-CS remain poorly defined.

This retrospective, multicenter, observational registry aims to evaluate the clinical outcomes and prognostic factors associated with mixed cardiogenic-vasoplegic shock. The study will analyze clinical, biological, and invasive hemodynamic data routinely collected during patient management for M-CS.

All included patients will have been admitted for cardiogenic shock, with or without vasoplegia, defined by low cardiac output and, when present, decreased systemic vascular resistance despite adequate filling pressures requiring vasopressor support.

The primary objective is to describe mortality and organ failure rates, while secondary analyses will identify determinants of adverse outcomes and potential phenotypic subgroups.

The PROMIX registry will be conducted across three French university hospitals (CHU Amiens-Picardie, CHU Dijon-Bourgogne, and CHU Rouen-Normandie).

This study is non-interventional, involving only data obtained as part of routine critical care, and will provide the first multicenter overview of this complex and underrecognized form of cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years old)
* Admitted to an intensive care unit for cardiogenic shock, at least SCAI stage C
* No opposition to data use

Exclusion Criteria:

* Missing key data, particularly regarding vasopressor doses and outcomes.
* Pregnant women
* Non-eligible shock etiologies, including but not limited to:
* Anaphylactic shock,
* Isolated hemorrhagic shock,
* Severe burns or major trauma,
* Severe acute pancreatitis,
* Fulminant hepatic failure,
* Neurogenic shock.
* Adult under legal protection (guardianship, curatorship, or judicial protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients (>18 years old) admitted to an intensive care unit for mixed cardiogenic shock (M-CS), defined by the coexistence of low cardiac output and, when present, vasoplegia requiring vasopressor support (norepinephrine >0.15 µg/kg/min) despite adequate filling pressures. Eligible patients must meet at least SCAI stage B criteria for cardiogenic shock.
  Patients with major missing data, particularly on vasopressor dosing, or those who have expressed opposition to data use will be excluded. This population represents a heterogeneous, high-risk group combining features of cardiogenic and vasoplegic circulatory failure, including ischemic, post-cardiotomy, and septic cardiomyopathy etiologies. The PROMIX study aims to better characterize clinical trajectories, hemodynamic profiles, and outcomes of these patients through clustering and phenotypic analyses.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 90 days | 90 days
  documented death occurring within 90 days following ICU admission

SECONDARY OUTCOMES:
Clinical characteristics and management trajectories | 90 days
  This outcome is descriptive in nature and aims to characterize the study population. Baseline variables (e.g., age, sex, cardiovascular history, comorbidities, and etiology of shock) will be reported separately using appropriate units for each variable (e.g., years, proportions, or categories), without aggregation into a single summary measure.
Phenotyping Cardiogenic Shock by Clustering | 90 days
  Identification of subgroups using unsupervised classification methods (clustering) and comparison of 90-day mortality rates.
Evolution of the SCAI Classification | 90 days
  Dynamic Evolution of the SCAI Classification (A to E) during the ICU stay. Each stage of classification is recording each day and during all ICU stay.
Evolution of Arterial Pressure | 7 days
  To assess the dynamic evolution of systolic, diastolic, and mean blood pressure (in mmHg) from Day 0 (D0) to Day 7 (D7)
Evolution of Norepinephrine Equivalent (NEE) Requirement | 7 days
  NEE (expressed in µg/kg/min) will be calculated at predefined time points: D0, D1, D3, D5, and D7, using standardized conversion factors to express all vasopressor doses as norepinephrine equivalents.
Evolution of Vasopressor Requirement | 7 days
  To assess the dynamic evolution of vasopressor and inotropic support quantified using the Vasopressor-Inotropic Score (VIS).
  VIS is calculated as a composite score based on standardized doses of vasopressors and inotropes, with higher scores indicating greater vasopressor and inotropic support (worse hemodynamic severity).
  VIS values will be assessed at predefined time points Day 0, Day 1, Day 3, Day 5, and Day 7 after shock onset.
Clinical outcomes | 90 days
  Use of renal replacement therapy and mechanical circulatory support (VA-ECMO, Impella, intra-aortic balloon pump).
ICU length of stay | 90 days
  Duration of ICU length of stay (days) since the ICU admission
Hospital lenght of stay | 90 days
  Duration of the Hospital lenght of stay (days) since the hospital admission and home discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Somme, France

IPD SHARING:
Plan to Share IPD: No